CLINICAL TRIAL: NCT04140136
Title: The Efficacy and Safety of Vitamin E Mixed Tocotrienols In Patients With Amyotrophic Lateral Sclerosis (ALS) : A Pilot Exploratory Study
Brief Title: The Efficacy and Safety of Vitamin E Mixed Tocotrienols In Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Professor Nortina Shahrizaila, Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018613-6392
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): This is a pilot randomized, double-blind, placebo-controlled, parallel-group study to evaluate the effects of 24-weeks tocotrienols (Tocovid Suprabio) supplementation in ALS patients.The investigational product is to be administered twice daily, at a dose of 400mg per day.
  Interventions: Dietary Supplement: Tocotrienols
- Placebo group (Placebo Comparator): This is a pilot randomized, double-blind, placebo-controlled, parallel-group study to evaluate the effects of 24-weeks tocotrienols (Tocovid Suprabio) supplementation in ALS patients. The placebo is similar in appearance but does not contain tocotrienols and consist of palm oil.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienols — Tocotrienols as a potent antioxidant to modulate oxidative stress and inflammatory response
  Arms: Treatment group
Dietary Supplement: Placebo — The placebo is similar in appearance, but does not contain tocotrienols and consist of palm oil
  Arms: Placebo group

SUMMARY:
There is currently no effective treatment in ALS. Oxidative stress, probably interacting with other neurodegenerative processes, is hypothesized to play a leading role in pathogenesis. These include mechanisms that promote glutamate excitotoxicity, mitochondrial dysfunction and axonal dysfunction.

In a transgenic mouse model of fALS that develops a disease with a clinical phenotype similar to ALS, dietary vitamin E supplementation delayed disease onset and slowed progression, although it did not prolong survival. When used as an experimental therapy in human trials, vitamin E did not affect survival significantly, but possibly slowed ALS progression. Two large, prospective epidemiologic studies suggest that longterm use of vitamin E supplements could be inversely associated with risk of ALS or ALS death. In another study, higher baseline serum α-tocopherol was associated with lower subsequent risk of ALS. A modest, non-significant protective effect from supplementation was seen in subjects with baseline serum α-tocopherol levels below median levels. In the current study, we aim to investigate the effects of tocotrienols in patients with ALS, particularly in delaying disease progression as well as assessing its safety profile in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a decrease of 1 to 4 points on the ALSFRS-R score during the 12-weeks observation period prior to screening and enrollment
* Patients of less than 2 years after the diagnosis of ALS.
* Patients without respiratory symptoms (orthopnea, dyspnea)
* Capable of giving signed informed consent

Exclusion Criteria:

* Patients who have developed respiratory failure necessitating ventilation
* Patients who have developed unsafe swallowing necessitating enteral feeding tube insertion
* Patients with other neurodegenerative disease such as Parkinson's disease and significant mental health illness
* Patients with certain concomitant diseases which may affect the assessment of safety/efficacy i.e. malignancy within the last 5 years, congestive heart disease, liver disease, kidney failure, bleeding disorders and other autoimmune diseases etc.
* Pregnant, lactating, and probably pregnant patients.
* Patients taking vitamin E tocopherol or tocotrienols supplements within 1 month from screening and randomisation.
* Patients who have participated in other trials within 12 weeks before consent, or who are participating in other clinical trials at present.
* Women of child bearing potential or nursing mother, unless they are willing to practice effective contraceptive measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean change of revised ALS Functional Rating Scale (ALSFRS-R) at baseline and 6 months between treatment group difference. | 6 months
  Efficacy of oral mixed Tocotrienols in patients with ALS in delaying disease progression as assess based on the cumulative score of ALSFRS-R between treatment group difference at specific time point.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events,haematological,renal and liver profile monitored at every visit | 6 months
  Safety of oral mixed Tocotrienols in ALS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Investigation Centre (CIC), Kuala Lumpur, Malaysia